CLINICAL TRIAL: NCT07350317
Title: A Non-Inferiority Randomized Controlled Trial Comparing Subcutaneous Natural Progesterone (Prolutex) vs. Cetrorelix Acetate for Luteinizing Hormone Surge Suppression in Freeze-All IVF Cycles.
Brief Title: Trial Comparing Subcutaneous Natural Progesterone (Prolutex) vs. Cetrorelix Acetate for Luteinizing Hormone Surge Suppression in Freeze-All IVF Cycles.
Acronym: IVF ART
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Trust Fertility Clinic (Other)
Responsible Party: Principal Investigator, ahmed Elbohoty, professor consultant ART, Trust Fertility Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BH/REC/149/25
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Assisted Reproductive Techniques
Keywords: ivf protocol; prolutex; premature ovulation
MeSH Terms: interventions — Control Groups; cetrorelix

STUDY DESIGN:
Intervention Model Description: * Design: Prospective, Phase IV, randomized, open-label, non-inferiority trial
  * Setting: Trust Fertility Clinic, Abu Dhabi, UAE
  * Randomization: 1:1 block randomization, stratified by age and ovarian reserve
  * Arms:
    * Control Group (A): Cetrorelix acetate 0.25 mg Subcutaneously daily from day 5 to trigger
    * Test Group (B): Natural progesterone 25 mg Subcutaneously (Prolutex) daily from day 5 to trigger
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (A): (Other): Cetrorelix acetate
  Interventions: Drug: Control Group (A):
- Test Group (B): (Experimental): Natural progesterone 25 mg Subcutaneously (Prolutex) daily from day 5 to trigger
  Interventions: Drug: Test Group (B):

INTERVENTIONS:
Drug: Control Group (A): — Control Group (A): Cetrorelix acetate 0.25 mg Subcutaneously daily from day 5 to trigger
  Other Names: Cetrorelix acetate 0.25 mg Subcutaneously daily from day 5 to trigger o
  Arms: Control Group (A):
Drug: Test Group (B): — prolutex
  Other Names: Natural progesterone 25 mg Subcutaneously (Prolutex) daily from day 5 to trigger
  Arms: Test Group (B):

SUMMARY:
The prevention of premature luteinizing hormone (LH) surge during controlled ovarian stimulation (COS) is critical for optimizing outcomes in assisted reproductive technology (ART). Cetrorelix acetate, a GnRH (Gonadotropin releasing hormone) antagonist administered subcutaneously, is the current standard for luteinizing hormone suppression. However, natural progesterone in a novel subcutaneous formulation (Prolutex) may offer a viable alternative.

Prolutex is a water-soluble complex of natural progesterone with hydroxypropyl-β-cyclodextrin (HPBCD), patented as US Patent No. 4,727,064 Pitha, Jallowing for subcutaneous injection. This may simplify treatment and improve patient compliance.

Progesterone forms are well studied and used globally/in UAE to suppress Luteinizing Hormone surge. It is an example of off-label use, which becomes a standard indication for use of progesterone. Several studies have demonstrated that exogenous progesterone can effectively suppress Luteinizing Hormone release while maintaining follicular development and oocyte competence. Furthermore, progestin-based protocols are potentially more cost-effective and similar to administer compared to GnRH (Gonadotropin releasing hormone) antagonists.

To our knowledge, this is the first randomized trial directly comparing a subcutaneous progesterone formulation (Prolutex) with cetrorelix acetate, administered via the same route, in terms of luteinizing hormone surge suppression. For this specific research, there are no relevant published studies available. This Randomised controlled trial will be done to address the research gap and compare the two already approved standard of care medications to see if Prolutex can be used as a viable alternative to suppress Luteinizing Hormone levels.

DETAILED DESCRIPTION:
Title: A Non-Inferiority Randomized Controlled Trial Comparing Subcutaneous Natural Progesterone (Prolutex) vs. Cetrorelix Acetate for Luteinizing Hormone Surge Suppression in Freeze-All IVF Cycles.

1. Principal Investigator:

   Prof. Ahmed Elbohoty, MSc, MD, FRCOG, EFRM Trust Fertility Clinic, Abu Dhabi, UAE Email: ahmed.elbohoty@trustfertility.com

   Co-Investigators:

   Dr Walid Sayed - Group Medical Director Trust Fertility Clinic Dr Irfan Aslam - Group IVF Lab director Trust Fertility Clinic Dr Amani Kanan - Specialist Obstetrics and Gynaecology Dr Nayrouz Gezaf - Specialist Obstetrics and Gynaecology Study Registration: To be registered on ClinicalTrials.gov Ethics Approval: To be approved by the Institutional Review Board (IRB) of Burjeel Holdings

   Standard IVF Procedures Under Institutional Coverage:

   All procedures-ovarian stimulation, hormone monitoring, and oocyte retrieval-are identical to routine clinical practice already being conducted at Trust fertility clinic - Burjeel Medical City.

   Participants will receive the same monitoring and safety precautions as standard IVF patients.

   No additional interventions will be introduced, and all clinical care will remain within the framework of the institution's established protocols.

   Both the investigators and the institution are covered under existing malpractice and liability insurance policies, which apply to all routine fertility procedures.

   Ethical Safeguards in Place:

   Participants will provide detailed informed consent, outlining all aspects of the protocol, including the use of approved medications and the lack of deviation from standard care.
2. Background: The prevention of premature luteinizing hormone (LH) surge during controlled ovarian stimulation (COS) is critical for optimizing outcomes in assisted reproductive technology (ART). Cetrorelix acetate, a GnRH (Gonadotropin releasing hormone) antagonist administered subcutaneously, is the current standard for luteinizing hormone suppression. However, natural progesterone in a novel subcutaneous formulation (Prolutex) may offer a viable alternative.

   Prolutex is a water-soluble complex of natural progesterone with hydroxypropyl-β-cyclodextrin (HPBCD), patented as US Patent No. 4,727,064 (Pitha, J.), allowing for subcutaneous injection. This may simplify treatment and improve patient compliance.

   Progesterone forms are well studied and used globally/in UAE to suppress Luteinizing Hormone surge. It is an example of off-label use, which becomes a standard indication for use of progesterone. Several studies have demonstrated that exogenous progesterone can effectively suppress Luteinizing Hormone release while maintaining follicular development and oocyte competence. Furthermore, progestin-based protocols are potentially more cost-effective and similar to administer compared to GnRH (Gonadotropin releasing hormone) antagonists.

   To our knowledge, this is the first randomized trial directly comparing a subcutaneous progesterone formulation (Prolutex) with cetrorelix acetate, administered via the same route, in terms of luteinizing hormone surge suppression. For this specific research, there are no relevant published studies available. This Randomised controlled trial will be done to address the research gap and compare the two already approved standard of care medications to see if Prolutex can be used as a viable alternative to suppress Luteinizing Hormone levels.

   Study Objectives:

   Primary Objective:

   To evaluate whether subcutaneous natural progesterone (Prolutex) is non-inferior to Cetrorelix Acetate in preventing premature ovulation in freeze-all IVF cycles.
3. Secondary Objectives:

   To compare the number of retrieved oocytes, MII rate, fertilization rate, and blastocyst formation rate To assess duration of ovarian stimulation To monitor hormone levels (luteinizing hormone, estradiol, progesterone) To evaluate patient tolerability, comfort, and adherence To compare cost-effectiveness of both protocols

   Study Design:

   Design: Prospective, Phase IV, randomized, open-label, non-inferiority trial Setting: Trust Fertility Clinic, Abu Dhabi, UAE Randomization: 1:1 block randomization, stratified by age and ovarian reserve

   Arms:

   Control Group (A): Cetrorelix acetate 0.25 mg Subcutaneously daily from day 5 to trigger Test Group (B): Natural progesterone 25 mg Subcutaneously (Prolutex) daily from day 5 to trigger
4. Sample Size Justification:

   Based on previous studies, the incidence of premature ovulation in GnRH (Gonadotropin releasing hormone) antagonist cycles is ~5% (Griesinger et al., 2016; Vuong et al., 2021). A non-inferiority margin of 5% (i.e., 10% total threshold) is selected, aligned with clinical tolerance standards (Fatemi et al., 2019). With α = 0.05 (one-sided) and 80% power, the minimum sample required is 102 per group. Allowing for a 10% dropout, the total enrolment target is 230 participants (115 per group).

   Data will be populated in excel and the data collection form will be attached to the participant file and upload to the secure study database.
5. Eligibility Criteria:

   Inclusion Criteria:

   Women aged 18-40 years Body Mass Index < 35 kg/m² Antral Follicle Count ≥ 8 or Anti-Müllerian Hormone ≥ 1.2 ng/mL Undergoing freeze-all IVF (for Ovarian Hyperstimulation Syndrome - OHSS risk, PGT- Preimplantation Genetic Testing, or personal preference)

   Exclusion Criteria:

   Poor responders (Bologna criteria) Stage III-IV endometriosis Pituitary or hypothalamic dysfunction Planned fresh embryo transfer Severe Male Factor. Semen Count <1 ×〖10〗^6 (<1 Million/ml) or Azoospermia)
6. Stimulation Protocol:

   Stimulation:

   Ovarian stimulation will begin between Cycle Day 2 and Cycle Day 5 of spontaneous or withdrawal-induced menstruation, as determined by physician assessment and baseline ultrasound and hormonal evaluation.

   Ovarian stimulation will be performed using human menopausal gonadotropin (HMG) or recombinant FSH, based on physician discretion and patient characteristics.

   Starting dose (typically 150-300 IU daily) will be individualized based on age, BMI (body mass index), AMH (Anti Mullerian Hormone), and Antral Follicle Count The choice of gonadotropin will be documented, and distribution between study arms will be analyzed to ensure balance.

   LUTEINIZING HORMONE Suppression:

   Cetrorelix acetate 0.25 mg Subcutaneously (control) Natural progesterone 25 mg Subcutaneously (Prolutex) (intervention) Starting on stimulation day 5 until the day of ovulation trigger Trigger: Either Triptorelin 0.2 mg Subcutaneously or recombinant hCG (Human Chorionic Gonadotropin), per physician assessment Oocyte Retrieval: 36 hours post-trigger Embryo Handling: Blastocyst culture followed by vitrification for all embryos (with or without embryo biopsy)

   Standard IVF Procedures Under Institutional Coverage:

   All Procedures - ovarian stimulation, hormone monitoring, and oocyte retrieval - are identical to routine clinical practice already being conducted at Trust Fertility Clinic - Burjeel Medical City.

   Participants will receive the same monitoring and safety precautions as standard IVF patients.

   No additional interventions will be introduced, and all clinical care will remain within the framework of the institution's established protocols.

   The study treatment and assessments will be covered by patient medical insurance/self-pay as these are considered standards of care. There are no additional expected risks beyond what the participants would typically encounter in a standard IVF cycle, in which case patient will receive appropriate medical care from the hospital in line with their insurance/self-pay coverage.
7. Monitoring and Hormonal Assessment:

   Monitoring Schedule:

   Ultrasound folliculometry will be the primary tool for monitoring follicular development and detecting premature ovulation.

   Transvaginal ultrasound assessments will be performed on:

   Stimulation Day 5 Stimulation Day 8 Trigger Day

   Each scan will evaluate:

   Number and size of growing follicles Ovarian response to stimulation Signs of follicular rupture or collapse Presence of free fluid in the pouch of Douglas Serum Luteinizing Hormone, estradiol (E2), and progesterone (P4) will be measured on the same days for hormonal profiling.

   In the Prolutex group, elevated progesterone is expected due to exogenous administration and will not be used to define premature ovulation.

   Ultrasound-based folliculometry will serve as the primary diagnostic tool for premature ovulation. Serum Luteinizing Hormone levels will be recorded as supportive data only.
8. Safety Monitoring:

   Incidence and grading of OHSS- Ovarian Hyperstimulation Syndrome Local injection reactions Patients will be followed up for any side effects/ reactions or complications. All such cases will be reported to the Principal Investigator.

   Minimal Risk Profile:

   This is a Phase IV, investigator-initiated study involving two medications-Cetrorelix acetate and natural progesterone (Prolutex®)-both of which are:

   Licensed and widely used in routine clinical practice; Administered within their approved clinical indications for LH suppression and luteal support in IVF; Associated with a well-established safety profile, with no investigational or experimental compounds introduced.

   There are no additional risks to participants beyond what they would typically encounter in a standard IVF cycle.

   Not a First-in-Human or High-Risk Study:

   Cetrorelix is a widely used GnRH antagonist, and Prolutex® is a subcutaneous formulation of bioidentical progesterone, complexed with hydroxypropyl-β-cyclodextrin, and has been shown in multiple studies to be both effective and well-tolerated and even safer that oral synthetic progestins.

   This study does not involve dose escalation, novel administration techniques, or vulnerable populations. It is designed to compare two clinically accepted protocols, differing only in the agent used for LH suppression.
9. Interim Safety Analysis:

   An interim analysis will be performed after 40 participants are enrolled in each group. It will assess:

   Premature ovulation rate in Prolutex group Early safety concerns If the Prolutex group exhibits an ovulation rate above 10% or significantly higher than control, the trial may be terminated early for safety reasons.
10. Outcomes:

    Primary Outcome:

    Premature ovulation, defined by:

    Ultrasound evidence of follicular rupture, including:

    Disappearance or collapse of dominant follicles Appearance of free fluid in the posterior cul-de-sac Absence of expected follicular structures at the time of oocyte retrieval Serum Luteinizing Hormone ≥ 10 IU/L or a ≥ 3-fold rise from baseline may be recorded as supportive, but ultrasound findings will be the definitive diagnostic criterion.

    Secondary Outcomes:

    Number of oocytes retrieved MII oocyte rate Fertilization rate Blastocyst formation rate Duration of stimulation (in days) Hormonal profile (Luteinizing Hormone, Estradiol, Progesterone) OHSS (Ovarian Hyperstimulation Syndrome) incidence Patient satisfaction and tolerability Cost-effectiveness
11. Cost-Effectiveness Analysis:

    Cost-effectiveness will be analyzed from the healthcare provider perspective by calculating the direct medical cost per effective outcome, including:

    Cost Inputs:

    Medication (Prolutex or Cetrotide + gonadotropins) Monitoring (Ultrasound and labs) Trigger medication Management of OHSS (Ovarian Hyperstimulation Syndrome) or complications Ovum pick-up cost Fertilization cost Embryo monitoring cost

    Effectiveness Measures:

    Cost per MII oocyte Cost per blastocyst Cost per successful suppression of Luteinizing Hormone surge

    Metrics:

    Cost-Effectiveness Ratio (CER) = Total Cost ÷ Outcome Incremental Cost-Effectiveness Ratio (ICER) = (Cost₁ - Cost₂) ÷ (Effectiveness₁ - Effectiveness₂) Sensitivity analyses will assess the impact of pricing variability and ovulation rate differences.
12. Study Duration:

The estimated duration of this study is 9 months, including recruitment, interim analysis, and data completion. Each participant will undergo a single stimulation cycle lasting approximately 2 weeks. Interim analysis will be conducted after 80 participants complete the cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-40 years.
2. Body Mass Index < 35 kg/m²
3. Antral Follicle Count ≥ 8 or Anti-Müllerian Hormone ≥ 1.2 ng/mL
4. Undergoing freeze-all IVF (for Ovarian Hyperstimulation Syndrome - OHSS risk, PGT- Preimplantation Genetic Testing, or personal preference)

Exclusion Criteria:

1. Poor responders (Bologna criteria)
2. Stage III-IV endometriosis
3. Pituitary or hypothalamic dysfunction
4. Planned fresh embryo transfer
5. Severe Male Factor. Semen Count <1 ×〖10〗^6 (<1 Million/ml) or Azoospermia)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females undergoing ovarian stimulation
Enrollment: 230 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: | 2 weeks within administration
  Ultrasound evidence of follicular rupture, including:
  1. Disappearance or collapse of dominant follicles
  2. Appearance of free fluid in the posterior cul-de-sac3. Absence of expected follicular structure

SECONDARY OUTCOMES:
secondary outcomes | 2 weeks after stimulation
  Number of oocytes retrieved
maturation rate | 2 weeks after stimulation
  • MII oocyte rate
• Fertilization rate | 2 days after egg collection
  fertilized number of m2 injected oocystes
• Blastocyst formation rate | 3 weeks after stimulation
  number of embryos reaching blastocysts
• Duration of stimulation (in days) | 10 to 14 days from start
  duration of stimulation in days
• Hormonal profile (Luteinizing Hormone, Estradiol, Progesterone) | 2 weeks duration from start of stimulation
  numeric hormone level

IPD SHARING:
Plan to Share IPD: No
not decided yet

REFERENCES:
- [Background] 1. Griesinger G, et al. Reprod Biol Endocrinol. 2016;14(1):29 2. Fatemi HM, et al. Hum Reprod. 2019;34(7):1223-34 3. Vuong LN, et al. Fertil Steril. 2021;116(5):1148-57 4. Papanikolaou EG, et al. J Assist Reprod Genet. 2020;37(4):841-50 5. Pitha J. US Patent No. 4,727,064